CLINICAL TRIAL: NCT03458039
Title: Evaluating Implementation Strategies to Scale-up Transdiagnostic Evidence-based Mental Health Care in Zambia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Infectious Disease Research in Zambia (Other)
Collaborators: Johns Hopkins University (Other); University of Alabama at Birmingham (Other); Education Development Center, Inc. (Industry); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH115495 (NIH)
Record Dates: First submitted 2018-02-15; First posted 2018-03-08 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Depression; Post-traumatic Stress Disorder; Anxiety; Substance Abuse
Keywords: mental health capacity building; low and middle-income country; train the trainer strategy; technology-based training; implementation science; adolescents and young adults (AYA)
MeSH Terms: conditions — Depression; Stress Disorders, Post-Traumatic; Anxiety Disorders; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Adolescents and young adults (AYA) with indicated mental health or behavioral health problems will be randomized to either the in-person CETA (n = 150), T-CETA (n=150), or treatment as usual condition (n = 100), for a total of 400 AYA participants. Each counselor will be trained in both CETA and T-CETA delivery methods.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the trainings, masking of AYA participants is not possible. Outcomes assessors who evaluate counselor competency will be masked to the randomization scheme. Data analysts will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- In-person CETA (Experimental): This is the in-person delivery method of the Common Elements Treatment Approach (CETA).
  Interventions: Behavioral: In-person CETA
- Telephone CETA (T-CETA) (Experimental): This is the technology-based delivery method for the Common Elements Treatment Approach (CETA).
  Interventions: Behavioral: Telephone CETA
- Treatment As Usual (Active Comparator): This is the treatment as usual control condition who will engage with their usual care in the community and will receive CETA, if desired, following completion of the study.
  Interventions: Behavioral: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: In-person CETA — The Common Elements Treatment Approach (CETA) is a transdiagnostic, multi-problem intervention designed to address adult and youth trauma, depression, anxiety, safety, and substance use. It is comprised of a small set of common elements found to be efficacious and prevalent across a range of EBTs to treat common mental health problems. CETA was designed to be flexible in the elements utilized, their order, and their dose (number of sessions) to allow counselors to address heterogeneity, comorbidity, and symptom fluctuations in and across clients. Treatment typically consists of 6 to 12 weekly, approximately 60-minute sessions delivered by lay workers.
  Other Names: CETA
  Arms: In-person CETA
Behavioral: Telephone CETA — For adaptation of the CETA manual for telephone delivery, the Applied Mental Health Research (AMHR) Group at Johns Hopkins University (JHU) reviewed evidence-based telehealth strategies and recommendations, telehealth ethical and legal guidelines, and clinical recommendations from telehealth providers. In addition, local TTTs in multiple contexts reviewed telehealth modifications and provided input that was incorporated into the final T-CETA manual used in this study. No changes were made to the structure, duration, and dose of CETA sessions, treatment components, or measurement-based clinical decision-making processes. Telehealth modifications, additions, and strategies were incorporated throughout the manual in delineated "telehealth boxes." This way, the original manual was maintained outside of the telehealth boxes, allowing for clear identification and training of telehealth modifications for both new and existing CETA counselors.
  Other Names: T-CETA
  Arms: Telephone CETA (T-CETA)
Behavioral: Treatment as Usual (TAU) — The control condition is defined as 'treatment as usual'. In Zambia, there are no formal services or standard of care treatments for mental and behavioral health problems among AYA. There are, however, organizations (such as non-governmental organizations) operating in Lusaka that provide intermittent services for these types of problems. Some AYA receive informal counseling from parish priests or other leaders in their communities. In this study we are therefore defining these types of informal services as 'treatment-as-usual.' We will closely track the type, number, and degree of these kinds of services that all participants receive and access. Following the conclusion of the study, we will offer the CETA intervention to control participants if it has been found to be safe and effective
  Other Names: TAU
  Arms: Treatment As Usual

SUMMARY:
This study utilizes a Hybrid Type 1 multi-arm parallel group randomized control design to compare the effectiveness of an evidence-based treatment (CETA) delivered either in-person or via telephone, compared with a treatment as usual (TAU) control group, on improving adolescent and young adult (AYA) mental and behavioral health outcomes. The study will also gather information on counselor treatment knowledge, fidelity and competency following a technology-delivered training. Lastly, the cost associated with these strategies will be explored to inform future scale-up of training and services. This study will be conducted in Lusaka, Zambia and participants will be enrolled at four different levels: prospective CETA trainers, prospective CETA counselors, AYA clients, and research/organizational staff. AYA clients are the primary participant type.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate implementation and service delivery strategies that can reduce the science-to-practice gap of evidence-based treatments (EBT) for mental health. Although evidence suggests that mental health treatments are acceptable and efficacious in low-and-middle income countries (LMIC) for the treatment of common mental disorders, there remains a gap in our understanding of how to bring these interventions to scale. Significant challenges include the high cost of in-person training, sustaining counselors in EBT, and limited client access to effective care.

The aim of this study is to test whether delivery of telephone CETA (T-CETA) can produce non-inferior, or similar, results to the standard in-person CETA for reducing mental and behavioral health problems among AYA and whether CETA and T-CETA are superior to treatment as usual (TAU) in reducing these problems. The study design is a randomized, non-inferiority trial. CETA trainers (up to n=6) will be identified from an existing cadre of Zambian trainers-in-training (TTT), who will facilitate technology-delivered trainings for prospective counselors (up to n = 50) from several partner organizations in Zambia. Counselors who participate in the training will be trained in both in-person CETA and T-CETA. Once trained, counselors will provide treatment to AYA clients randomized to the CETA or T-CETA condition. Following completion of the study, TAU control participants will be offered CETA.

The transdiagnostic treatment being scaled up, CETA, was effective in several previous randomized clinical trials in LMIC settings with lay providers, including in Zambia. CETA provides the basis for feasible scale-up through the use a single therapy to treat multiple common mental disorders with varying severities, an approach that is more cost-effective than implementing multiple single-disorder focused psychotherapy treatments in LMIC.

Primary outcomes will be AYA client mental health and behavioral health outcomes. Secondary outcomes include trainer and counselor CETA competency and knowledge, and qualitative interviews of the acceptability, appropriateness, feasibility, and scale-up potential of technology-based CETA training and treatment delivery. The cost-effectiveness of the technology training strategy and the two treatment delivery methods will also be evaluated.

The project will specifically strengthen the capacity of: 1) study staff to conduct mental health clinical science research, 2) counselor and trainers in CETA training, supervision and delivery, and 3) policy and decision makers to interpret and appropriately utilize the scientific evidence to improve mental health policies and programs. This proposal leverages previous studies and strong collaborations in Zambia with the Ministry of Health and numerous local organizations. Results from this trial will produce effectiveness and costing data on treatment delivery strategies that could inform the scale-up potential of diverse EBT in LMIC across and beyond mental health. This research study ultimately addresses both the treatment and implementation gaps in lower-resource settings globally.

ELIGIBILITY:
CETA Counselors

Inclusion:

1. 18 years of age or older
2. Interest in providing CETA
3. Time/availability to participate in the study
4. Minimal education level is comparable to a high school education
5. Ability to speak English fluently and speak at least 1 local language (Nyanja or Bemba)
6. Completion of an in-person interview with study team investigators demonstrating strong communication skills
7. Planning to stay in study area (Lusaka) to provide treatment to clients

Exclusion:

1. If previously trained in CETA

CETA Trainers

Inclusion:

1. All eligibility criteria for CETA counselors
2. Interest in teaching CETA
3. Completion of the CETA training
4. Completion of a minimum of 3 CETA cases under supervision

Adolescent/Young Adult (AYA) Clients

Inclusion:

1. 15-29 years of age
2. Attend or be referred to study site
3. Live in the area served by a study site (i.e., not staying temporarily)
4. Ability to speak one of the study languages (English, Bemba, or Nyanja)
5. Screening: Present with one or more common mental/behavioral health problems based on validated screening tools included in the audio computer assisted self-interviewing (ACASI) system. Specifically, the following screening tools and cut-off values:

   1. Youth Self Report Internalizing Scale (≥14)
   2. Youth Self Report Externalizing Scale (≥8)
   3. Child PTSD Symptom Scale (≥11.5)

Exclusion:

1. Currently on unstable psychiatric drug regimen (e.g., altered in past two months)
2. Suicide attempt or active and severe self-harm in past month
3. Psychotic disorder or severe mental illness

Research/Organizational Staff

Inclusion:

1. Involved in development and/or implementation of the technology training platform, including clinical, research, and web development staff.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change in adolescent and young adult (AYA) internalizing and externalizing symptoms as measured by the Youth Self Report | Baseline; within one month following CETA treatment (~3-4 months post-baseline for TAU participants); 6-month follow-up after treatment (~9 months post-baseline for TAU).
Change in adolescent and young adult (AYA) trauma symptoms as measured by the Child PTSD Symptom Scale | Baseline; within one month following CETA treatment (~3-4 months post-baseline for TAU participants); 6-month follow-up after treatment (~9 months post-baseline for TAU).

SECONDARY OUTCOMES:
Change in adolescent and young adult (AYA) substance use as measured by the ASSIST | Baseline; within one month following CETA treatment (~3-4 months post-baseline for TAU participants); 6-month follow-up after treatment (~9 months post-baseline for TAU).
Change in adolescent and young adult (AYA) physical health and functioning as measured by the EQ-5D-Y | Baseline; within one month following CETA treatment (~3-4 months post-baseline for TAU participants); 6-month follow-up after treatment (~9 months post-baseline for TAU).
Trainer competency & knowledge of Common Elements Treatment Approach (CETA). | Outcomes at the trainer level will be assessed at three time points: 1) after CETA counselor training (baseline), 2) three months into active cases (3 months post-baseline), and 3) at posttreatment (~9 months post-baseline).
  Assess competency and knowledge of trainers in training CETA using locally developed measures of competency and knowledge.
Counselor competency & knowledge of Common Elements Treatment Approach (CETA). | Outcomes at the counselor level will be assessed at three time points: 1) after baseline CETA counselor training, 2) three months into active cases (3 months from baseline), and 3) following provision of CETA treatment (~9 months post-baseline).
  Assess competency and knowledge of counselors in training CETA using locally developed measures of competency and knowledge.
Cost effectiveness of adapting training for technology delivery, and in-person and telephone delivery of CETA. | Costs assessed throughout course of the study up to 48 months.
  Cost-effectiveness analyses will calculate health utility values by deriving quality adjusted life years (QALYs) from health states reported at each follow up time point by AYA, and then estimate mean QALYs gained per treatment condition
Challenges, advantages, feasibility, acceptability, and sustainability of a technology-delivered training and supervision model. | Trainer and counselor qualitative interviews will be conducted at two time points: 1) After counselor training (baseline), and 2) At post-treatment of CETA cases (~9 months post-baseline).
  Qualitative interviews with trainers and counselors regarding technology training and treatment delivery strategies. Qualitative results will be used to support and enrich quantitative findings and to refine, support, and troubleshoot future iterations of technology-driven training.
Challenges, advantages, feasibility, acceptability, and sustainability of a telephone-delivered treatment delivery model (T-CETA). | AYA qualitative interviews will be conducted at CETA posttreatment (~3 months post-baseline).
  Qualitative interviews with AYA clients regarding technology treatment delivery strategies. Qualitative results will be used to support and enrich quantitative findings and to refine, support, and troubleshoot future iterations of technology-driven treatment provision.

CONTACTS AND LOCATIONS:
Overall Officials: Izukanji Sikazwe, MBChB, Principal Investigator — Chief Executive Officer
Locations (1):
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
All necessary steps will be taken to ensure adherence to all NIH guidelines on sharing raw data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Pending
Access Criteria: Pending
URL: http://www.cidrz.org

REFERENCES:
- [Background] Kieling C, Baker-Henningham H, Belfer M, Conti G, Ertem I, Omigbodun O, Rohde LA, Srinath S, Ulkuer N, Rahman A. Child and adolescent mental health worldwide: evidence for action. Lancet. 2011 Oct 22;378(9801):1515-25. doi: 10.1016/S0140-6736(11)60827-1. Epub 2011 Oct 16. PMID 22008427
- [Background] Benjet C. Childhood adversities of populations living in low-income countries: prevalence, characteristics, and mental health consequences. Curr Opin Psychiatry. 2010 Jul;23(4):356-62. doi: 10.1097/YCO.0b013e32833ad79b. PMID 20520546
- [Background] Saxena S, Thornicroft G, Knapp M, Whiteford H. Resources for mental health: scarcity, inequity, and inefficiency. Lancet. 2007 Sep 8;370(9590):878-89. doi: 10.1016/S0140-6736(07)61239-2. PMID 17804062
- [Background] Kakuma R, Minas H, van Ginneken N, Dal Poz MR, Desiraju K, Morris JE, Saxena S, Scheffler RM. Human resources for mental health care: current situation and strategies for action. Lancet. 2011 Nov 5;378(9803):1654-63. doi: 10.1016/S0140-6736(11)61093-3. Epub 2011 Oct 16. PMID 22008420
- [Background] Ray ML, Wilson MM, Wandersman A, Meyers DC, Katz J. Using a training-of-trainers approach and proactive technical assistance to bring evidence based programs to scale: an operationalization of the interactive systems framework's support system. Am J Community Psychol. 2012 Dec;50(3-4):415-27. doi: 10.1007/s10464-012-9526-6. PMID 22711269
- [Background] Pearce J, Mann MK, Jones C, van Buschbach S, Olff M, Bisson JI. The most effective way of delivering a train-the-trainers program: a systematic review. J Contin Educ Health Prof. 2012 Summer;32(3):215-226. doi: 10.1002/chp.21148. PMID 23173243
- [Background] Murray LK, Skavenski S, Kane JC, Mayeya J, Dorsey S, Cohen JA, Michalopoulos LT, Imasiku M, Bolton PA. Effectiveness of Trauma-Focused Cognitive Behavioral Therapy Among Trauma-Affected Children in Lusaka, Zambia: A Randomized Clinical Trial. JAMA Pediatr. 2015 Aug;169(8):761-9. doi: 10.1001/jamapediatrics.2015.0580. PMID 26111066
- [Derived] Figge CJ, Kane JC, Skavenski S, Haroz E, Mwenge M, Mulemba S, Aldridge LR, Vinikoor MJ, Sharma A, Inoue S, Paul R, Simenda F, Metz K, Bolton C, Kemp C, Bosomprah S, Sikazwe I, Murray LK. Comparative effectiveness of in-person vs. remote delivery of the Common Elements Treatment Approach for addressing mental and behavioral health problems among adolescents and young adults in Zambia: protocol of a three-arm randomized controlled trial. Trials. 2022 May 19;23(1):417. doi: 10.1186/s13063-022-06319-4. PMID 35590348